CLINICAL TRIAL: NCT02755051
Title: Targeting Sleep in Kids With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Christina McCrae, Principal Investigator, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004675
Record Dates: First submitted 2016-03-11; First posted 2016-04-28 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Autism Spectrum Disorder; Chronic Insomnia
MeSH Terms: conditions — Autism Spectrum Disorder; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBT-CI-A Therapy (Experimental): Participants in this group receive Cognitive Behavioral Therapy for children with Chronic Insomnia and Autism Spectrum Disorder (CBT-CI-A)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy for children with Chronic Insomnia and Autism Spectrum Disorder involves 8, one-hour sessions of a non-drug cognitive behavioral intervention. Session content listed below:
  1. Sleep education
  2. Sleep scheduling, limit setting, and stimulus control
  3. Teaching relaxation strategies and other adaptive coping skills
  4. Parenting strategies (differential attention, rewards, consequences)
  5. Identification of maladaptive & adaptive cognitions
  6. Problem solving & communication skills
  7. Sleep restriction; bright light to change circadian rhythms
  8. Review gains and plan for long-term maintenance
  Other Names: CBT-CI-A

SUMMARY:
Children with Autism Spectrum Disorder (ASD) and insomnia, and their parent(s) will undergo 8 sessions of Cognitive Behavioral Therapy designed for Children with Chronic Insomnia and ASD (CBT-CI-A). Treatment delivery will be assessed for each session. Treatment receipt will be assessed at the end of session 3. Treatment enactment will be assessed throughout treatment, post-treatment, and follow-up. Sleep and secondary outcomes (child daytime behavior, parent sleep) will be collected at baseline, post-treatment, and 1-month follow-up.

Study Flow:

Baseline (wk1-2) ---> CBT-CI-A (wk3-10) ---> Post-Treatment (wk11-12) --->Wks 13-16 --->Follow-up (wk 17-18)

Session:

1. Sleep education
2. Sleep scheduling, limit setting, and stimulus control
3. Teaching relaxation strategies and other adaptive coping skills
4. Parenting strategies (differential attention, rewards, consequences)
5. Identification of maladaptive & adaptive cognitions
6. Problem solving & communication skills
7. Sleep restriction; bright light to change circadian rhythms
8. Review gains and plan for long-term maintenance

DETAILED DESCRIPTION:
Children with ASD and insomnia, and their parent(s) will undergo 8 sessions of CBT-CI-A. Treatment delivery will be assessed for each session. Treatment receipt will be assessed at the end of session 3. Treatment enactment will be assessed throughout treatment, post-treatment, and follow-up. Sleep and secondary outcomes (child daytime behavior, parent sleep) will be collected at baseline, post-treatment, and 1-month follow-up.

Children (6-12 yrs; n = 30) who meet full DSM (Diagnostic and Statistical Manual) criteria18 for ASD and insomnia will be recruited from an existing clinical registry database. Eligibility criteria for initial recruitment will include IQ (intelligence quotient) of 75 or above (to ensure ability to participate in cognitive components of treatment), previous DSM diagnosis of ASD, and previous evaluation using gold standard diagnostic tools, including the Autism Diagnostic Observation Schedule (ADOS)27 and/or Autism Diagnostic Interview - Revised (ADI-R).28 The Thompson Center database currently includes 337 children with ASD ages 6-12 who have completed the ADOS and/or ADIR and have IQ>75. Following initial recruitment, eligibility for participation will include DSM diagnosis of insomnia. Insomnia will be diagnosed by study staff using gold standard diagnostic tools, a brief (10 min.) structured interview, Child Sleep Habits Questionnaire29, and sleep diaries.30 Child will report or parent will observe sleep latency (time to fall asleep) or wake during the night >30 minutes that is confirmed by baseline sleep diaries. Dr. Sahota will provide referrals for children with suspected sleep apnea. Additional criteria will include participation of the child's parent or legal guardian living in the same home, and parental ability to read and understand English at the 5th grade level. Given previous experience, size of the database and insomnia prevalence in ASD, the investigators expect no difficulty recruiting our target sample size.

Treatment will be manualized and individually administered by graduate students trained by Drs. McCrae and Mazurek. Parent and child will be actively involved in treatment.

CBT-CI-A will use established behavioral sleep strategies.5-7 Treatment will be adapted from a manualized protocol developed and tested by Dr. McCrae in TD children. Adaptations for children with ASD will be based on Dr. Mazurek's experience and expertise, practice pathway recommendations of the ATN, and previously published CBT adaptations for treatment of anxiety in children with ASD. Adaptations will include increased use of visual supports, greater opportunities for repetition/practice, incorporation of special interests, and video modeling.

ELIGIBILITY:
Inclusion Criteria:

* previous Diagnostic and Statistical Manual of Mental Disorders diagnosis of Autism Spectrum Disorder, and previous evaluation using gold standard diagnostic tools, including the Autism Diagnostic Observation Schedule (ADOS)27 and/or Autism Diagnostic Interview - Revised (ADI-R).
* Who have IQ>75.
* Child will report or parent will observe sleep latency (time to fall asleep) or wake during the night >30 minutes that is confirmed by baseline sleep diaries.
* Participation of the child's parent or legal guardian living in the same home, and parental ability to read and understand English at the 5th grade level.

Exclusion Criteria:

* unable to provide informed consent
* unable to implement treatment due to sleep disorder other than insomnia (i.e., sleep apnea [apnea/hypopnea index, AHI >15], Periodic Limb Movement Disorder (PLMD [myoclonus arousals per hour >15])
* bipolar or seizure disorder (due to risk of sleep restriction treatment)
* other major psychopathology except depression or anxiety (e.g., suicidal ideation/intent, psychotic disorders)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Subjective Sleep at 12 weeks | Daily for 12 weeks from Baseline thru Post-treatment
  With parental assistance, all child participants will complete daily sleep diaries each morning
Change from Baseline Objective Sleep at 12 weeks | Continuously for 2 weeks at Baseline and 2 weeks at Post-treatment
  Child participants will wear an actigraph all day for those weeks
Change from Baseline Subjective Sleep at 18 weeks | Daily 18 weeks from Baseline thru Follow-up
  With parental assistance, all child participants will complete daily sleep diaries each morning
Change from Baseline Objective Sleep at 18 weeks | Continuously for 2 weeks at Baseline, 2 weeks at Post-treatment and 2 weeks at Follow-up
  Child participants will wear an actigraph during those weeks

SECONDARY OUTCOMES:
Child Behavior at Baseline | To be completed at 2 weeks
  The Aberrant Behavior Checklist is a 58-item parent-report measure of daytime problem behaviors
Child Behavior at Post-treatment | To be completed at 12 weeks
  The Aberrant Behavior Checklist is a 58-item parent-report measure of daytime problem behaviors
Child Behavior at Follow-up | To be completed at 18 weeks
  The Aberrant Behavior Checklist is a 58-item parent-report measure of daytime problem behaviors
Change in subjective Parent Sleep from Baseline at 12 weeks | Daily for 12 weeks from Baseline thru Post-treatment
  Parents will complete daily sleep diaries each morning
Change in subjective Parent Sleep from Baseline at 18 weeks | Daily for 18 weeks from Baseline thru Follow-up
  Parents will complete daily sleep diaries each morning
Change in objective Parent Sleep from Baseline at 12 weeks | Continuously for 2 weeks at Baseline and 2 weeks at Post-treatment
  Parents will wear an actigraph during those weeks
Change in objective Parent Sleep from Baseline at 18 weeks | Continuously for 2 weeks at Baseline, 2 weeks at Post-treatment, and 2 weeks at Follow-up
  Parents will wear an actigraph during those weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christina S McCrae, Ph. D, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Department of Health Psychology, University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No